CLINICAL TRIAL: NCT06697743
Title: Post Bariatric Surgery Acute Kidney Injury: Incidence and Risk Factors
Status: Not yet recruiting | Type: Observational
Sponsor: Georgina Tharwat Abdelmasih (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Georgina Tharwat Abdelmasih, Dr Georgina Tharwat, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Post bariatric surgery AKI
Record Dates: First submitted 2024-11-14; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Bariatric Surgery; Acute Kidney Injury
Keywords: Bariatric surgery; Acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patient undergo bariatric surgery: 1. Inclusion criteria:
     1. Age more than 18 years old undergo bariatric surgery .
     2. BMI ≥30 : ( BMI = weight in kg / height in m²)
  2. Exclusion criteria:
     1. previous kidney diseases(AKI , CKD) .
     2. patients unfit for surgery e.g ( comorbidities : CHD , LCF ) 3. Drugs : (ACE-I , ARBs, and NSAIDS)

SUMMARY:
Bariatric surgery is the most effective means of inducing and maintaining sustained weight loss. Apart from the weight loss effect, bariatric surgery leads to the remission of chronic metabolic disorders such as type 2 diabetes (T2D) and hypertension . Recent studies have shown that bariatric surgery improves renal perfusion and glomerular function and reduces inflammatory markers which can lead to an improvement of microalbuminuria and proteinuria However, acute kidney injury (AKI) can complicate the postoperative course after bariatric surgery. The etiology of AKI after bariatric surgery can be multifactorial and complex in obese population . The preexisting factors such as diabetes, hypertension, and CKD in these patients can additionally worsen the renal insult during the postoperative period . Postoperative AKI is associated with increase morbidity and mortality especially in cases of severe AKI that requires dialysis support . Identifying the high-risk patients for development of postoperative AKI would prevent renal injury. Our aim was to study the incidence and etiology of postoperative AKI after bariatric surgery . Causes of post bariatric surgery AKI include . Pre renal causes :dehydration ( repeated vomiting and diarrhoea)which are common complications post bariatric surgery , haemorrhagic shock (from the site of anastomosis , ulcer ) , septic shock ( leakage , pneumonia) , hypotension and respiratory depression secondary to narcotic overdose. Rena causes: contract induced nephropathy after using CT scan guided drainage of intra abdominal collection post operative, Rhabdomylosis , drug induced nephropathy e.g :using of IV vancomycin for sepsis in ICU .. many causes can lead to AkI post bariatric surgery but the common two causes are dehydration and sepsis .

ELIGIBILITY:
1. Inclusion criteria:

   1. Age more than 18 years old undergo bariatric surgery .
   2. BMI ≥30 : ( BMI = weight in kg / height in m²)
2. Exclusion criteria:

   1. previous kidney diseases(AKI , CKD) .
   2. patients unfit for surgery e.g ( comorbidities : CHD , LCF ) 3. Drugs : (ACE-I , ARBs, and NSAIDS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: multi central study in Egypt
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
incidence | Baseline
  assess the incidence of postoperative AKI after bariatric surgery .
Risk factors | Baseline
  assess the risk factors of postoperative AKI after bariatric surgery

SECONDARY OUTCOMES:
duration of hospitalization | Baseline
  Assess the duration of hospitalization, and it's relation with the incidence of AKI
readmission | Baseline
  Assess the duration of readmission within 30 d after surgery and it's relation with the incidence of AKI

REFERENCES:
- [Background] Inker LA, Eneanya ND, Coresh J, Tighiouart H, Wang D, Sang Y, Crews DC, Doria A, Estrella MM, Froissart M, Grams ME, Greene T, Grubb A, Gudnason V, Gutierrez OM, Kalil R, Karger AB, Mauer M, Navis G, Nelson RG, Poggio ED, Rodby R, Rossing P, Rule AD, Selvin E, Seegmiller JC, Shlipak MG, Torres VE, Yang W, Ballew SH, Couture SJ, Powe NR, Levey AS; Chronic Kidney Disease Epidemiology Collaboration. New Creatinine- and Cystatin C-Based Equations to Estimate GFR without Race. N Engl J Med. 2021 Nov 4;385(19):1737-1749. doi: 10.1056/NEJMoa2102953. Epub 2021 Sep 23. PMID 34554658
- [Background] Levin A, Ahmed SB, Carrero JJ, Foster B, Francis A, Hall RK, Herrington WG, Hill G, Inker LA, Kazancioglu R, Lamb E, Lin P, Madero M, McIntyre N, Morrow K, Roberts G, Sabanayagam D, Schaeffner E, Shlipak M, Shroff R, Tangri N, Thanachayanont T, Ulasi I, Wong G, Yang CW, Zhang L, Robinson KA, Wilson L, Wilson RF, Kasiske BL, Cheung M, Earley A, Stevens PE. Executive summary of the KDIGO 2024 Clinical Practice Guideline for the Evaluation and Management of Chronic Kidney Disease: known knowns and known unknowns. Kidney Int. 2024 Apr;105(4):684-701. doi: 10.1016/j.kint.2023.10.016. PMID 38519239
- [Background] Morgan DJ, Ho KM. Acute kidney injury in bariatric surgery patients requiring intensive care admission: a state-wide, multicenter, cohort study. Surg Obes Relat Dis. 2015 Nov-Dec;11(6):1300-6. doi: 10.1016/j.soard.2015.01.005. Epub 2015 Jan 14. PMID 25892347
- [Background] Huang H, Lu J, Dai X, Li Z, Zhu L, Zhu S, Wu L. Improvement of Renal Function After Bariatric Surgery: a Systematic Review and Meta-analysis. Obes Surg. 2021 Oct;31(10):4470-4484. doi: 10.1007/s11695-021-05630-4. Epub 2021 Aug 6. PMID 34355340
- [Background] Lee Y, Anvari S, Chu MM, Lovrics O, Khondker A, Malhan R, Aditya I, Doumouras AG, Walsh M, Hong D. Improvement of kidney function in patients with chronic kidney disease and severe obesity after bariatric surgery: A systematic review and meta-analysis. Nephrology (Carlton). 2022 Jan;27(1):44-56. doi: 10.1111/nep.13958. Epub 2021 Aug 16. PMID 34375462
- [Background] Wilhelm SM, Young J, Kale-Pradhan PB. Effect of bariatric surgery on hypertension: a meta-analysis. Ann Pharmacother. 2014 Jun;48(6):674-82. doi: 10.1177/1060028014529260. Epub 2014 Mar 24. PMID 24662112
- [Background] Moriconi D, Manca ML, Anselmino M, Rebelos E, Bellini R, Taddei S, Ferrannini E, Nannipieri M. Predictors of type 2 diabetes relapse after Roux-en-Y Gastric Bypass: A ten-year follow-up study. Diabetes Metab. 2022 Jan;48(1):101282. doi: 10.1016/j.diabet.2021.101282. Epub 2021 Sep 18. PMID 34547450